CLINICAL TRIAL: NCT05576844
Title: Developing and Validating a Sleep Promotion Intervention Program for People Living With HIV Based on Social Rhythm Theory
Brief Title: Ai Youmian (Love Better Sleep) for People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Jingjing MENG, PhD candidate, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021zzts0334; CX20210113 (Other Grant/Funding Number: The Hunan Provincial Innovation Foundation for Postgraduate)
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Sleep; HIV Infections
Keywords: social rhythm; sleep quality; people living with HIV
MeSH Terms: conditions — HIV Infections; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal and social rhythm intervention (Experimental)
  Interventions: Behavioral: 8-week interpersonal and social rhythm intervention
- Controlled group (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: 8-week interpersonal and social rhythm intervention — The development of the intervention strategies are based on social rhythm theory, interpersonal and social rhythm therapy, and previous research results, and the intervention aims to improve sleep by stabilizing participants' social rhythm and increasing the amount of interpersonal communication.
  Arms: Interpersonal and social rhythm intervention
Other: Usual care — Control group participants received usual care, including daily disease management and routine drug guidance.
  Arms: Controlled group

SUMMARY:
People living with HIV (PLWH) frequently report sleep disturbances. The social rhythm theory, which proposes that stressful life events can interfere with sleep by disrupting the stability of daily routines, provides new insights into identifying predictors of sleep disturbances and improving sleep in PLWH. This study is a randomized controlled trial. PLWH with poor self-reported sleep quality (Pittsburgh sleep quality index>7) was randomly divided into a control group or an intervention group. The control group receives the usual care, that is, daily disease management and routine drug guidance (set as waitlist). The intervention group received a sleep promotion intervention program based on social rhythm theory, along with daily disease management and routine drug guidance. The intervention period was 8 weeks, once a week, and the duration of each intervention was about 40-60 minutes. The sleep-related outcome indicators were measured before the intervention (T0), immediately after the intervention (T1), and 3 months after the intervention (T2), and the participants' social rhythm, daytime sleepiness, sleep belief and attitude, depression, etc. were evaluated to verify the effects of the intervention. At the same time, participants who insisted on completing all intervention modules were selected from the intervention group after the end of the whole study. Self-designed satisfaction questionnaires and semi-structured interviews were used to understand the participants' experience and feedback on the intervention program. In addition, the investigator asked the reasons for the withdrawal of participants who withdrew from the study through an interview during the outcome period.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection,
2. Aged 18 years or above,
3. Total score of Pittsburgh sleep quality index > 7,
4. Possess basic literacy,
5. Voluntary participation in the study.

Exclusion Criteria:

1. Self reported previous diagnoses of severe sleep disorder disorders such as obstructive sleep apnea, restless legs syndrome, periodic limb movement of sleep, nocturnal urinary frequency or diurnal phase shift disorder,
2. Initiation of antiretroviral therapy within the past 30 days or change in antiretroviral therapy regimen within the past 30 days,
3. Current treatment with psychotropic medication, or use of any medication with sedative or excitatory effects,
4. Working in jobs that require night shifts that may affect the circadian rhythm and no consideration of changing jobs in the recent month,
5. Currently participating in other research projects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
change of sleep quality | Outcomes was evaluated before the intervention (T0), after the 8-week intervention (T1), and 3 months follow-up after the intervention (T2)
  Pittsburgh sleep quality index (PSQI) was used. The scale consists of 18 items divided into 7 dimensions. Each dimension is scored from 0 to 3. The total PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality.

SECONDARY OUTCOMES:
change of social rhythm | Outcomes was evaluated before the intervention (T0), after the 8-week intervention (T1), and 3 months follow-up after the intervention (T2)
  The Brief Social Rhythm Scale was used. The scale consists of 10 items to assess the regularity of daily activities during the week. The regularity of each activity is rated on a 6-point Likert type scale. The total BSRS score ranges from 10 to 60, with higher total scores reflecting greater irregularity of the daily activities.
change of sleepiness | Outcomes was evaluated before the intervention (T0), after the 8-week intervention (T1), and 3 months follow-up after the intervention (T2)
  The Epworth Sleepiness Scale was used. It contains 8 questions, each scoring 0-3 with increasing number signifying higher chance of "dozing" while engaged in specific activities of daily life.
change of sleep beliefs and attitudes | Outcomes was evaluated before the intervention (T0), after the 8-week intervention (T1), and 3 months follow-up after the intervention (T2)
  The Dysfunctional Beliefs and Attitudes about Sleep was used. The scale consists of 16 items. The scoring range for each item was from 1 to 5 and the sum of scores of all 16 items ranged from 16 to 80. The lower total score indicates the more erroneous beliefs a participant has.
change of coping styles | Outcomes was evaluated before the intervention (T0), after the 8-week intervention (T1), and 3 months follow-up after the intervention (T2)
  Simplified Coping Style Questionnaire was used. The 20-item scale includes 2 dimensions, positive coping (12 items) and negative coping (8 items). Each item is scored on a 4-point Likert scale, with higher scores indicating greater positive/negative coping styles. The mean scores for the positive and negative items were the final scores for positive and negative coping, respectively.
change of social support | Outcomes was evaluated before the intervention (T0), after the 8-week intervention (T1), and 3 months follow-up after the intervention (T2)
  Perceived Social Support Scale was used. The 12-item scale uses a 7-point Likert scale, with total scores ranging from 12 to 84, with higher scores indicating higher levels of perceived social support.
change of depression symptoms | Outcomes was evaluated before the intervention (T0), after the 8-week intervention (T1), and 3 months follow-up after the intervention (T2)
  The self-rating depression scale was used. The scale included 20 items and each item was scored on a 4-point Likert scale to examine the frequency of the occurrence of assessed depression symptoms over the previous week. The total raw score ranged from 20 to 80, with higher scores indicating higher levels of depression symptoms.
change of interpersonal competence | Outcomes was evaluated before the intervention (T0), after the 8-week intervention (T1), and 3 months follow-up after the intervention (T2)
  Interpersonal Competence Questionnaire was used. The scale included 40 items and each item was scored on a 5-point Likert scale. The total score ranged from 40 to 200, with higher scores indicating higher levels of interpersonal competence.

OTHER OUTCOMES:
sleep diary | Participants in the intervention group were required to record a sleep diary after getting up on a daily basis during the 8-week intervention, which was used to guide adjustment of the weekly intervention strategy.
  Bedtime, sleep latency, times of waking up during the night, self-rated sleep quality, time of getting up in the morning, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing MENG, Principal Investigator — Central South University
Locations (1):
- The First Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The participants in this study were all HIV/AIDS patients. Due to sexual and HIV-related stigma and discrimination, HIV/AIDS patients are reluctant to inform others of their infection status. At recruitment, participants were also informed that the data were anonymous and presented in a total sample format to help alleviate their reluctance and concerns about privacy breaches.

REFERENCES:
- [Background] Wu J, Wu H, Lu C, Guo L, Li P. Self-reported sleep disturbances in HIV-infected people: a meta-analysis of prevalence and moderators. Sleep Med. 2015 Aug;16(8):901-7. doi: 10.1016/j.sleep.2015.03.027. Epub 2015 May 18. PMID 26188954
- [Background] Ning CX, Chen XX, Lin HJ, Qiao XT, Xu YY, Shen WW, Zhao D, He N, Ding YY. [Characteristics of sleep disorder in HIV positive and HIV negative individuals: a cluster analysis]. Zhonghua Liu Xing Bing Xue Za Zhi. 2019 May 10;40(5):499-504. doi: 10.3760/cma.j.issn.0254-6450.2019.05.002. Chinese. PMID 31177727
- [Background] Lee KA, Gay C, Portillo CJ, Coggins T, Davis H, Pullinger CR, Aouizerat BE. Types of sleep problems in adults living with HIV/AIDS. J Clin Sleep Med. 2012 Feb 15;8(1):67-75. doi: 10.5664/jcsm.1666. PMID 22334812
- [Background] Pujasari H, Chung MH. Sleep Disturbance in the Context of HIV: A Concept Analysis. SAGE Open Nurs. 2022 Apr 20;8:23779608221094541. doi: 10.1177/23779608221094541. eCollection 2022 Jan-Dec. PMID 35493547
- [Background] Voss JG, Barroso J, Wang T. A Critical Review of Symptom Management Nursing Science on HIV-Related Fatigue and Sleep Disturbance. Int J Environ Res Public Health. 2021 Oct 12;18(20):10685. doi: 10.3390/ijerph182010685. PMID 34682431
- [Background] Grandin LD, Alloy LB, Abramson LY. The social zeitgeber theory, circadian rhythms, and mood disorders: review and evaluation. Clin Psychol Rev. 2006 Oct;26(6):679-94. doi: 10.1016/j.cpr.2006.07.001. Epub 2006 Aug 10. PMID 16904251
- [Background] Monk TH, Reynolds CF 3rd, Buysse DJ, DeGrazia JM, Kupfer DJ. The relationship between lifestyle regularity and subjective sleep quality. Chronobiol Int. 2003 Jan;20(1):97-107. doi: 10.1081/cbi-120017812. PMID 12638693
- [Background] Haynes PL, Kelly M, Warner L, Quan SF, Krakow B, Bootzin RR. Cognitive Behavioral Social Rhythm Group Therapy for Veterans with posttraumatic stress disorder, depression, and sleep disturbance: Results from an open trial. J Affect Disord. 2016 Mar 1;192:234-43. doi: 10.1016/j.jad.2015.12.012. Epub 2015 Dec 24. PMID 26748739